CLINICAL TRIAL: NCT02490189
Title: Comparative Trial of a Mindfulness-based Intervention Versus Cognitive Behavior Therapy for Social Anxiety Disorder
Brief Title: Mindfulness-based Intervention Versus CBT for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); University of Ottawa (Other)
Responsible Party: Principal Investigator, Diana Koszycki, Professor and Research Chair in Mental Health, Hopital Montfort
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK-27-02-15
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention (Experimental): Participants in the mindfulness-based intervention arm will receive 12 weekly sessions of 2 to 2.5 hours duration. The intervention will be delivered in a group format. Participants will be assigned weekly homework.
  Interventions: Behavioral: Mindfulness-based Intervention
- Cognitive Behavior Group Therapy (Active Comparator): Participants in the cognitive behavior group therapy arm will receive 12 weekly sessions of 2 to 2.5 hours in duration. Participants will be assigned weekly homework.
  Interventions: Behavioral: Cognitive Behavior Group Therapy

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — Twelve week group intervention that includes training in mindfulness meditation, self-compassion and mindful exposure.
  Arms: Mindfulness-Based Intervention
Behavioral: Cognitive Behavior Group Therapy — Twelve week group intervention that focuses on the interaction between thoughts, feelings, and behaviors.
  Other Names: CBGT
  Arms: Cognitive Behavior Group Therapy

SUMMARY:
To conduct a prospective, randomized trial to compare the efficacy of a group mindfulness-based intervention adapted for social anxiety disorder (MBI-SAD) versus cognitive behavior group therapy (CBGT).

DETAILED DESCRIPTION:
The main aim of this comparative trial is to determine if the MBI-SAD will be noninferior to CBGT in improving core symptoms of social anxiety disorder, depressive symptoms, self, esteem, disability and quality of life. A secondary aim is to examine whether treatment gains are maintained over a 6-month period. Exploratory aims of the study are to: 1) determine if the MBI-SAD enhances self-compassion and mindfulness relative to CBGT; 2) determine if changes in self-compassion and mindfulness mediate the clinical response to the MBI-SAD; and 3) explore moderators of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of social anxiety disorder (SAD) of at least moderate severity
* Montgomery Asberg Depression Rating Scale score ≤ 25
* Comorbid depressive disorders, panic disorder, agoraphobia, generalized anxiety disorder, specific phobias, eating disorders are allowed as long as the SAD is primary and predominates the clinical picture.

Exclusion Criteria:

* Coexisting Axis I disorders excluding those listed in the inclusion criteria
* Coexisting medical conditions that can alter the clinical presentation of SAD (e.g. Parkinson's disease)
* Lifetime history of bipolar disorder or psychotic symptoms
* Substance-related disorders in the last 12 months
* Acutely suicidal or history of suicide attempt in the past five years
* History of non-suicidal self-injurious behavior in the last 12 months
* Currently receiving psychotherapy
* Currently engaged in a regular meditation or yoga practice
* Unable to attend weekly group sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-07-25 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | Change from baseline to week 12 and 6-month follow-up
  A 24-item clinician-rated scale that assesses fear and avoidance of social performance and social situations.

SECONDARY OUTCOMES:
Social Phobia Inventory | Change from baseline to week 12 and 6-month follow-up
  A 17-item self-report scale that assesses symptom domains of social anxiety.
Clinical Global Impression Improvement Ratings | Change from baseline to week 12 and 6-month follow-up
  A 7-point clinician-rated scale that assesses level of clinical improvement.
Beck Depression Inventory | Change from baseline to week 12 and 6-month-follow-up
  A 21-item self-report measure of severity of depressive symptoms.
Social Adjustment Scale-Self Report Revised | Change from baseline to week 12 and 6-month follow-up
  A 49-item self-report scale that assesses functional impairment in multiple roles.
Rosenberg Self-Esteem Scale | Change from baseline to week 12 and 6-month follow-up
  A 10-item self-report measure of self-esteem.
Satisfaction with Life Questionnaire | Change from baseline to week 12 and 6-month follow-up
  A 5-item self-report scale that assesses overall satisfaction with life.

OTHER OUTCOMES:
Self-Compassion Scale-Short Form | Change from baseline to week 12 and 6-month follow-up
  A 12-item self-report scale that captures how respondents perceive their actions towards themselves in difficult times.
Five-Facet Mindfulness Questionnaire | Change from baseline to week 12 and 6-month follow-up
  A 39-item self-report inventory that assesses different facets of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Koszycki, PhD, Principal Investigator — Hopital Montfort
Locations (2):
- Canada (2):
  - Hopital Montfort, Ottawa, Ontario
  - Montfort Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No